CLINICAL TRIAL: NCT07006688
Title: A Phase 1, Multicenter, Open-Label, Safety and Pharmacokinetic Study of Orally Administered Ivosidenib in Participants With IDH1-Mutated Malignancies and Hepatic or Renal Impairment
Brief Title: A Study of an IDH1m Inhibitor in Participants With IDH1-Mutated Malignancies and Hepatic or Renal Impairment
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Servier Bio-Innovation LLC (Industry)
Collaborators: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S095031-218; 2024-517923-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: IDH1-Mutated Malignancies
MeSH Terms: interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 - Moderate Hepatic Impairment (HI) (Experimental)
  Interventions: Drug: Ivosidenib Oral Tablet
- Group 2 - Severe HI (Experimental)
  Interventions: Drug: Ivosidenib Oral Tablet
- Group 3 - Severe Renal Impairment (RI) (Experimental)
  Interventions: Drug: Ivosidenib Oral Tablet
- Group 4 - Adequate hepatic function (Experimental)
  Interventions: Drug: Ivosidenib Oral Tablet
- Group 5 - Adequate renal function (Experimental)
  Interventions: Drug: Ivosidenib Oral Tablet

INTERVENTIONS:
Drug: Ivosidenib Oral Tablet — 500mg Ivosidenib taken orally once daily for continuous 28-day cycles

SUMMARY:
The objective of this study is to investigate the PK, PD, safety, and tolerability of ivosidenib in adult participants with IDH1-mutated malignancies and hepatic impairment (HI)/ renal impairment (RI). Participants will be enrolled into one of 5 groups based on their hepatic or renal function. During the treatment period participants will have study visits on days 1, 4, 8, 15, 22, and 28 of Cycle 1, on days 1 and 15 of Cycle 2 and 3, and on day 1 of each additional cycle. Each cycle is 28 consecutive days of treatment and cycles will be continuous until the end of the study. Approximately 30 days after treatment has ended, a safety follow-up visit will occur. Study visits may include blood tests, ECG, vital signs, and a physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Participants with hematologic malignancies (including but not limited to acute myeloid leukemia (AML), myelodysplastic syndrome (MDS), myeloproliferative neoplasms, clonal cytopenia of unknown significance with a high-risk score [CHRS ≥12.5], chronic myelomonocytic leukemia, multiple myeloma, and non-Hodgkin's lymphoma) or solid tumors excluding glioma, with a locally confirmed IDH1 R132 mutation before Cycle 1 Day 1.
* Based on renal and hepatic function, participants within the:

  a. Moderate HI group, must have: i. Total bilirubin >1.5 to 3 × upper limit of normal (ULN), not linked to Gilbert's disease, and any aspartate aminotransferase (AST) value, ii. Adequate renal function as evidenced by creatinine clearance (CrCl) ≥60 mL/min estimated according to the Cockcroft-Gault formula. b. Severe HI group, must have: i. Total bilirubin >3 × ULN and any AST value, ii. Adequate renal function as evidenced by CrCl

  ≥60 mL/min estimated according to the Cockcroft-Gault formula. c. Severe RI group, must have: i. CrCl ≥15 to 29 mL/min estimated according to the Cockcroft-Gault formula, ii. Adequate hepatic function as evidenced by:
  1. Blood total bilirubin ≤1.5 × ULN, unless due to Gilbert's disease, where participants should have blood total bilirubin ≤3 × ULN;
  2. AST, alanine aminotransferase, and alkaline phosphatase ≤3.0 × ULN
* Participants of the control groups with adequate hepatic or renal function characterized as:

  1. Hepatic control group: Adequate hepatic function as evidenced by total bilirubin and AST ≤ULN, and normal to mild RI (CrCl ≥60 mL/min estimated according to the Cockcroft-Gault formula).
  2. Renal control group: Adequate renal function as evidenced by CrCl ≥90 mL/min (estimated according to the Cockcroft-Gault formula) and normal to mild HI (total bilirubin ≤1.5 × ULN, participants with Gilbert's disease should have blood total bilirubin ≤3 × ULN).
* Participants previously or currently treated with ivosidenib are eligible if treated at the 500 mg QD dose or if treated at the 250 mg QD dose due to strong cytochrome P450 (CYP)3A4 inhibitor intake. Participants with a hematologic malignancy on co-treatment with azacitidine are also eligible.
* WOCBP must agree to abstain from sexual intercourse or use 2 effective methods of birth control (a highly effective method and a barrier method) from the time of giving informed consent throughout the study and for 90 days after the last dose of ivosidenib. Hormonal contraception alone is not considered an acceptable method of contraception and should be combined with a barrier method.

Exclusion Criteria:

* Have undergone hematopoietic stem cell transplant (HSCT) within 60 days of the first dose of ivosidenib, or on immunosuppressive therapy post-HSCT at the time of screening, or with active acute or chronic graft-versus-host-disease (GVHD) requiring systemic therapy. (Participants with GVHD managed by minimal interventions [a physiologic dose of steroids] are permitted with the medical monitor's approval.)
* Have received systemic anticancer therapy (with the exception of azacitidine), investigational agent treatment, or radiotherapy <14 days, or had surgery <4 weeks before planned Cycle 1 Day 1 of ivosidenib, and/or did not recover from the AEs associated with these therapies and/or surgeries. In addition, the first dose of ivosidenib should not occur before a period of ≥5 half-lives of the study drug has elapsed.
* Have hematological diseases (other than AML or MDS) or solid tumors that are eligible for other treatments known to provide clinical benefit.
* Have received calcineurin inhibitors within 4 weeks prior to enrollment.
* Have significant active cardiac disease within 6 months before the start of ivosidenib, including NYHA Class III or IV congestive heart failure, myocardial infarction, unstable angina, and/or stroke.
* Use of any medications that are known to prolong the QT interval unless they can be transferred to other medications within ≥5 half-lives before dosing or unless the medications can be properly monitored during the study. (If equivalent medication is not available, QTcF should be closely monitored).
* Planned use of any strong CYP3A4 inducer or sensitive CYP3A4 substrate with a narrow therapeutic window or certain antifungals that are CYP3A4 substrates while the participant is receiving ivosidenib. Participants who are taking these medications must have the minimum washout period of ≥5 half-lives before the first dose of ivosidenib and not take the medications for the duration of their participation in the study.
* Have known active inflammatory gastrointestinal disease, chronic diarrhea, previous gastric resection or laparoscopic gastric banding, short-gut syndrome, gastroparesis, or other active conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally. Gastroesophageal reflux disease under medical treatment is allowed (assuming no drug interaction potential).
* Have a known familial history of sudden death or polymorphic ventricular arrhythmia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Maximum observed steady-state concentration (Cmax,ss) | Through day 28 of cycle 1
Area under the concentration time curve from 0 to 24 hours (AUC0-24hr) | Through day 28 of cycle 1
Predose plasma concentration (Ctrough) | Through day 28 of cycle 1
Time to maximum observed concentration (Tmax) | Through day 28 of cycle 1

SECONDARY OUTCOMES:
Area under the effect concentration-time curve from time point 0 (predose) up to 8 hours postdose (AUEC0-8hr) | Through day 28 of cycle 1
Percent inhibition for AUEC0-8hr (%BAUEC0-8hr) | Through day 28 of cycle 1
Single dose ivosidenib plasma concentrations, maximum observed concentration (Cmax) | Through day 28 of cycle 1
Single dose ivosidenib plasma concentrations AUC0-24hr | Through day 28 of cycle 1
Single dose ivosidenib plasma concentrations Tmax | Through day 28 of cycle 1
Steady-state unbound ivosidenib Cmax | Day 28 of cycle 1
Steady-state unbound ivosidenib Ctrough | Day 28 of cycle 1
Steady-state unbound ivosidenib AUC0-24hr | Day 28 of cycle 1
Number of Adverse Events (AEs) | Through the Safety Follow-up Visit, 30 days after last dose (approximately 3 years)
Number of Serious Adverse Events (SAEs) | Through the Safety Follow-up Visit, 30 days after last dose (approximately 3 years)
Number of Adverse Events of Special Interest (AESIs) | Through the Safety Follow-up Visit, 30 days after last dose (approximately 3 years)
Number of AEs leading to discontinuation | Through the Safety Follow-up Visit, 30 days after last dose (approximately 3 years)

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (2):
  - Icon Cancer Centre, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo, Brazil
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - START - Hospital HM Nou Delfos, Barcelona
  - START Madrid - Fundacion Jimenez Diaz, Madrid
  - START Madrid Centro Oncologico Clara Campal Sanchinarro Univesrity Hospital, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorization in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com/